CLINICAL TRIAL: NCT05520905
Title: Evaluation of the Feasibility, Acceptability, and Effectiveness of TelePrEP for At-risk Youth in Colorado
Brief Title: TelePrEP for At-risk Youth in Colorado
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-0588
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Hiv
Keywords: youth; telemedicine; telehealth; HIV; prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemedicine for pre-exposure prophylaxis of HIV (Experimental): 1. We will identify youth potentially eligibile for PrEP using tenfovir alefenamide/emtricitabine (TAF/FTC).
  2. Eligible youth will be contacted for rapid (same day) consenting and enrollment.
  3. Participants who consent to the study will undergo a PrEP initiation visit either the same day or within two weeks with a provider. The initial visit may be in-person or via Telemedicine.
  4. TelePrEP visits may be carried out in the setting of the participant's choosing and may include home or at a community organization.
  5. Recommended laboratory testing will be arranged as part of the PrEP initiation visit. HIV testing will be carried out as well as Centers for Disease Control and Prevention (CDC)-recommended laboratory testing will be obtained.
  6. TelePrEP(or in-person visits as needed) will be conducted by a skilled multidisciplinary team one month after initiation and then every three months.
  Interventions: Other: TelePrEP

INTERVENTIONS:
Other: TelePrEP — HIV pre-exposure prophylaxis delivered via telemedicine.

SUMMARY:
Youth represent the largest proportion of new HIV infections in Colorado, reflective of their inadequate access and uptake of pre-exposure prophylaxis(PrEP)for HIV prevention. Colorado's 2019 HIV/AIDS Prevention Program state-wide review of PrEP barriers showed PrEP eligible individuals do not access PrEP services due to lack of interest, not wanting referral to a navigator, and low estimation of HIV risk. The overall goal is to provide youth at higher risk for HIV with an effective youth informed telemedicine delivery of PrEP (TelePrEP) that addresses PrEP barriers and contributes to ending the HIV epidemic in Colorado. The primary objective will be proportion of youth retained on PrEP 12 months after initiation. The hypotheses are that a TelePrEP model for youth will be acceptable and feasible and will result in successful initiation, persistence and retention on oral PrEP.

ELIGIBILITY:
Inclusion Criteria:

* HIV negative
* Eligible for PrEP using emtricitabine (F)/tenofovir alafenamide (TAF) (F/TAF) (brand name Descovy) based on current CDC guidance
* assigned male at birth
* has had male sex partners in the past 6 months (and not in a monogamous partnership with a recently tested, HIV-negative man) and
* either any sex without a condom in the past 6 months or
* a bacterial sexually transmitted infection
* Consents to TelePrEPvisits
* Willing to use current insurance coverage for clinic and laboratory services OR willing to be assisted to obtain insurance coverage OR eligible for other coverage such as Title X funds or charity care

Exclusion Criteria:

* HIV-infection or concern for acute HIV infection until ruled out
* Pregnancy
* Persons at risk through receptive vaginal sex including cisgender women and transgender men (persons assigned female sex at birth)
* Persons with only injection drug indications for PrEP without sexual risk indications outlined in inclusion criteria

Ages: 14 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Retention | 48 weeks
  Retention on PrEP at week 48. Retention in PrEP care 12 months after initiation as defined by either PrEP clinic visit (telehealth or in-person) or prescription refill.

SECONDARY OUTCOMES:
TelePrEP Feasibility | 48 weeks
  Feasibility will be measured by 1) proportion of those screened and eligible who are initiated on PrEP, 2) persistence (time to first discontinuation), and 3) survey responses from participants identifying barriers and facilitators of TelePrEP (satisfaction survey).
TelePrEP Acceptability | 48 weeks
  Acceptability will be measured by 1) proportion who obtain PrEP services via TelePrEPfor at least 2 visits in a 12 month period and 2) electronic questionnaire responses from youth screening for PrEP at study enrollment as well as satisfaction surveys

OTHER OUTCOMES:
Uptake TelePrEP | 48 weeks
  Number (median; interquartile range) of TelePrEP visits carried out successfully with youth PrEP users by referral or initiation setting
TelePrEP visit rate | 48 weeks
  Number (median; interquartile range) of TelePrEP visits per patient in 12 month period vs. in-person visits per participant and associate patients demographics related to higher number of TelePrEP visits.
TelePrEP Satisfaction | 48 weeks
  PrEP user and provider satisfaction with TelePrEP services.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No